CLINICAL TRIAL: NCT05171803
Title: Investigating Immune Escape by SARS-CoV-2 Variants
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Advarra (Industry)
Responsible Party: Principal Investigator, Noah Kojima, MD, Principal Investigator, University of California, Los Angeles
Other Study IDs: PTL-2021-0007
Record Dates: First submitted 2021-12-16; First posted 2021-12-29 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; Immunity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention, prospective, cohort study.

SUMMARY:
The purpose of this protocol is to investigate the ability of pre-existing immunity by natural infection or vaccination to prevent infections by emerging SARS-CoV-2 variants.

DETAILED DESCRIPTION:
Several variants of the SARS-CoV-2 virus were identified in 2020 including the United Kingdom variant (known as 20I/501Y.V1, VOC 202012/01, or B.1.1.7), South Africa variant (known as 20H/501Y.V2 or B.1.35), and Brazil variant (known as P.1), with more variants still being discovered. There is concern that these variants, due to mutations in spike protein and receptor-binding domain of the spike protein, can be more infectious, lethal, and potentially escape the immune responses from vaccination or prior infection. Research is needed to understand the risks associated with currently known variants of SARS-CoV-2 as well as investigate if there is potential for new mutations to form that would allow SARS-CoV-2 variants to partially or entirely escape the immune mechanisms developed from vaccination and/or prior infection from the wild-type strain of SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* People who have been fully vaccinated for COVID-19 2-12 weeks prior to enrollment or individuals <3 months post-COVID-19 infection.
* Collection of samples for blood samples will be done only from healthy, nonpregnant adults who weigh at least 110 pounds.
* Participants must be able to provide informed consent.

Exclusion Criteria:

-Subjects considered vulnerable including children, pregnant women, nursing home residents, or other institutionalized persons, fetuses, prisoners, and persons without decisional capacity.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults living in Los Angeles County
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-05-29 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Assessing immunity | 1 year
  Assess immune escape among people with vaccination or natural immunity

CONTACTS AND LOCATIONS:
Locations (1):
- Curative, San Dimas, California, United States

IPD SHARING:
Plan to Share IPD: No
This will not be available.